CLINICAL TRIAL: NCT06930846
Title: HOBSCOTCH-CA (HOme-Based Self-management and COgnitive Training CHanges Lives in Brain CAncer)
Acronym: HOBSCOTCH-CA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Mayo Clinic (Other); University of North Carolina (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Elaine T. Kiriakopoulos, MD, MPH, MSc Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002841
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Brain Cancer; Brain Tumor; Brain Neoplasms; Primary Brain Tumor; Low-grade Glioma; Oligodendroglioma; Meningioma; Low Grade Astrocytoma; Cognitive Dysfunction; Memory Impairment; Memory Disorders; Memory Dysfunction
Keywords: Brain cancer survivor; Brain tumor survivor; Cognition; Self-management; Cognitive training; Memory disorders; Cognitive remediation; Caregiver; Caregiver burden; Mindfulness
MeSH Terms: conditions — Brain Neoplasms; Oligodendroglioma; Meningioma; Cognitive Dysfunction; Memory Disorders; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Waitlist Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CA Participant-Group 1 (Experimental): After enrollment and completion of baseline assessments, CA Participant Group 1 will receive the HOBSCOTCH-PTE intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions (option to do on webcam)
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: HOBSCOTCH-CA
- CA Participant-Group 2 (Active Comparator): After a 3-month waiting period and having completed baseline and 3-month study assessments, CA Participant Group 2 will receive the HOBSCOTCH-CA intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions (option to do on webcam)
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: HOBSCOTCH-CA
- CA Participant Caregiver-Group 1 (Experimental): After enrollment and completion of baseline assessments, CA Participant Caregiver Group 1 will receive an adapted version of HOBSCOTCH-CA alongside the CA participant by attending:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: HOBSCOTCH-CA
- CA Participant Caregiver-Group 2 (Active Comparator): After a 3-month waiting period and having completed baseline and 3-month study assessments, CA Participant Caregiver Group 2 will receive an adapted version of HOBSCOTCH-CA alongside the CA participant by attending:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: HOBSCOTCH-CA

INTERVENTIONS:
Behavioral: HOBSCOTCH-CA — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-CA is an adaptation of the HOBSCOTCH program for people who are survivors of brain cancer or a brain tumor that incorporates education about the effects from brain cancer/tumor and its treatment on cognition into the education module and gives them the option of enrolling with a Caregiver. CA Participants receive all sessions of HOBSCOTCH-CA. If they enroll with a Caregiver, the Caregiver participates in the education (introductory) session and sessions 1 and 8. The HOBSCOTCH-CA Participant may invite their Caregiver to attend all sessions.
  Other Names: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH)

SUMMARY:
The purpose of this study is to assess the ability of the home-based intervention, HOBSCOTCH-CA, to improve the quality of life and cognitive function in Service Members, Veterans and civilians who are survivors of brain cancer or a brain tumor (CA participants). This study will also assess the ability of the HOBSCOTCH-CA program to improve quality of life in caregivers of patients with brain cancer/tumor and to reduce caregiver burden. Enrolling with a Caregiver is optional for CA participants.

Investigators will compare two groups of CA participants and their Caregiver (enrolling with a Caregiver is optional): one who receives HOBSCOCTCH-CA immediately (Group 1) and another group that will receive HOBSCOTCH-CA (Group 2) after a 3-month waiting period. Participants will be in the study for about 6 months total.

HOBSCOTCH-CA involves 45 to 60 minute one on one virtual sessions with a certified Cognitive Coach including a "pre" program session and 8 weekly sessions thereafter. Participants will learn about problem solving therapy and mindfulness or relaxation training. CA participants are asked to do short homework assignments and keep a brief daily diary on a smart phone app. All participants complete study questionnaires or surveys at enrollment, 3 months later and at 6 months (at the end of the study).

DETAILED DESCRIPTION:
The investigators' hypothesis is that the home-based intervention (HOBSCOTCH-CA) will improve quality of life and cognitive function in Service Members, Veterans and civilians with who are survivors of brain cancer or tumor. Also, that the integration of family caregiver participation in the HOBSCOTCH-CA intervention will reduce caregiver burden and increase caregiver knowledge of their loved one's disease and the cognitive challenges they face, ultimately leading to an improvement in caregiver quality of life (QOL).

The investigators will test the hypothesis by pursuing the following specific aims:

Aim 1: Adapt the HOBSCOTCH program education module for delivery to patients with brain cancer/tumor (CA participant) and cognitive challenges.

The investigators' working hypothesis is that the existing education module of the HOBSCOTCH program can be adapted to address key knowledge areas for patients with brain cancer/tumor and their caregivers.

Aim 2: Evaluate the efficacy of the HOBSCOTCH-CA program in patients with brain cancer/tumor.

The investigators' working hypothesis is that the HOBSCOTCH-CA intervention will improve quality of life (QOL) in CA participants. The investigators also expect to see improvements in subjective cognition, knowledge, self-efficacy, symptom reduction, and health outcomes.

Aim 3: Incorporate family caregivers into select components of the HOBSCOTCH-CA intervention and evaluate the effects of the HOBSCOTCH-CA intervention on the caregiver.

The investigator's working hypothesis is that family caregivers will have improvement in QOL and reduced caregiver burden and improved health status as a result of their family member with CA participating in the HOBSCOTCH-CA intervention, and by their own participation in the HOBSCOTCH-CA modules delivering disease specific education and mindfulness skill building exercises.

ELIGIBILITY:
CA Participants will be referred to the study by their providers (Oncologist) who will be made aware of the study and inclusion/exclusion criteria. Inclusion Criteria 2. - 5. and Exclusion Criteria 1. - 3. will be confirmed by referring providers. Participants who learn about the study here and elsewhere will be instructed on how to confirm their eligibility with their provider.

Inclusion Criteria for CA Participant:

1. 18 + years
2. Service members, Veterans and civilians with a diagnosis of brain cancer (excluding glioblastoma)
3. Diagnosis of primary brain tumor with expected survival of 2 years or greater (e.g., low-grade glioma, oligodendroglioma, IDH mutant astrocytoma, meningioma) defined as the presence of a primary lesion on neuroimaging (CT or MRI), confirmed by histopathological examination (Note: some patients being treated for meningioma may be treated with radiotherapy without need for initial histopathologic confirmation)
4. Patients undergoing surgical and/or radiation therapy will have completed their treatment at least 3 months prior to being enrolled in trial (Note: patients receiving chemotherapy or other systemic therapy will be included)
5. Stable on all CNS acting medications for one month prior to enrollment
6. Subjective cognitive complaints
7. Literate and proficient in English
8. Internet access for the pre-session and Session 1 of the HOBSCOTCH-CA program; telephone access for sessions 2-8

Exclusion Criteria for CA Participant:

1. Presence of a neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease)
2. Acute psychiatric disorder or substance abuse
3. Patients with glioblastoma (GBM)

Inclusion Criteria for CA Participant Caregiver:

1. Age 18 +
2. Caregiver to a patient with a confirmed diagnosis of brain cancer/tumor survivor
3. CA Subject has given permission for their caregiver to participate
4. Literate and proficient in English
5. Internet access (for Pre-HOBSCOTCH and Session 1)
6. Telephone access (for Session 8)

Exclusion Criteria for CA Participant Caregiver:

1. Significant visual impairment precluding reading or writing
2. No reliable telephone or internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by comparing Neuro-QOL scores at baseline and at 3 months post-intervention in CA Participants. | Baseline and 3 months post-intervention
  The Neuro-QOL is a self-reported, validated assessment on health-related quality of life covering 17 domains in individuals with neurological disorders. Items are scored on a 5-point Likert scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. Depending on the domain, a higher or lower score can indicate better or poorer quality of life for that domain.
Change in quality of life as measured by comparing FACT-Br scores at baseline and at 3 months post-intervention in CA Participants. | Baseline and 3 months post-intervention
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is a validated instrument measuring general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 scales or domains. A 5-point Likert scale from 0 (not at all) to 4 (very much) is utilized with a higher score representing poorer or better QOL depending on the domain.
Change in subjective cognitive function as measured by comparing scores on the Cognitive Function Sub-Scale (Item Bank 2.0) of the Neuro-QOL at baseline and at 3 months post-intervention in CA Participants. | Baseline and 3 months post-intervention
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Change in CA Participant Caregiver burden as measured by comparing Zarit Burden Interview scores at baseline and at 3 months post-intervention in Caregivers of CA Participants. | Baseline and 3 months post-intervention
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5 point Likert scale is used with a higher score indicating a greater level of perceived burden.

SECONDARY OUTCOMES:
Changes in CA Participant knowledge of relationship between their condition and cognition and memory as measured by comparing scores on the HOBSCOTCH-CA Knowledge Questionnaire at baseline and at 6 months (end of study) | Baseline and at 6 months (at the end of the study).
Changes in CA Participants' objective cognition as measured by comparing scores on the Montreal Cognitive Assessment (MoCA) at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Montreal Cognitive Assessment (MOCA) is a validated 30 item test that helps healthcare professionals detect cognitive impairments. The test examines seven domains (aspects) of cognitive function with a total of 11 different exercises and tasks including: executive and visuospatial function, naming, attention, language, abstraction, delayed recall, orientation. Scores range from 0 - 30 with higher scores indicating less cognitive impairment.
Changes in CA Participants' subjective cognition as measured by comparing scores on the Everyday Memory Questionnaire (EMQ) at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Everyday Memory Questionnaire (EMQ) is a validated assessment that was developed as a subjective measure of memory failure in everyday life. It is composed of 13 items, with a Likert-type scale ranging from "once or less in the last month" (1) to "once or more once per day" (5); higher values indicate the presence of subjective memory complaints.
Changes in CA participants' executive function as measured by comparing scores on the self-reported Behavior Inventory of Executive Function-Adult Version (BRIEF-A) at baseline and 3-months post intervention. | Baseline and 3 months post-intervention
  The BRIEF-A is a standardized measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment that includes 75 items within nine scales of executive function. All 75 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). Raw scores for each scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores indicate greater impairment in executive functioning.
Changes in CA participants' self-efficacy as measured by comparing scores on the PROMIS (Patient-Reported Outcomes Measurement Information System) Item Bank v1.0 General Self-Efficacy assessment at baseline and 3-months post-intervention. | Baseline and 3 months post-intervention
  The PROMIS self-efficacy scales is a validated measure designed to assess an individual's confidence in managing various situations, problems and events. 10 items are self-reported on a scale of 1 (I am not at all confident) to 5 (I am very confident). Lower scores indicate poorer perception of self-efficacy.
Changes in CA Participants' mood as measured by comparing scores on the Patient Health Questionnaire (PHQ-9) at baseline and at 3 months post- intervention. | Baseline and 3 months post-intervention
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria on a 4-point Likert scale as "0" (not at all) to "3" (nearly every day). Higher scores are consistent with greater symptoms of poor mood or depression.
Changes in CA participants' anxiety as measured by comparing score on the Generalized Anxiety Disorder-7 (GAD-7) at baseline and at 3-months post-intervention. | Baseline and 3 months post-intervention
  The Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring symptoms of generalized anxiety disorder (GAD). The seven items are scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Higher scores suggest greater symptoms of anxiety.
Changes in CA participants' symptom frequency as measured by a daily self-reported diary compared at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  CA participants will self-report symptoms related to their brain cancer/tumor using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in CA participants' medication adherence as measured by a daily self-reported diary compared at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  CA participants will self-report their medication adherence activity using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in CA participants' use of memory strategies as measured by a daily self-reported diary compared at baseline and 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  CA participants will self-report their use of the memory strategies they learn in the HOBSCOTCH-CA program using a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in a paper log.
Changes in CA participants' self-reports of wellbeing as measured by comparing daily reports of well-being in a diary at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention.
  The researchers will collect daily well-being information throughout the entire study by use of a smartphone app or paper log and a basic single item Likert-scale of well-being.
Engagement and Satisfaction for CA Participants as measured by analyzing study attrition and a Participant Satisfaction Survey at the end of the study. | At 6 months (end of the study).
  The Participant Satisfaction Survey has been developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It contains 10 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program. Participants also have the option to write open text about their experiences in the HOBSCOTCH-CA intervention.
Engagement and Satisfaction for CA Participants as measured by CollaboRATE post-study completion. | At 6 months (end of the study).
  CollaboRATE is a brief, 3 item patient-reported measure of shared decision making, namely the perception of being informed and then involved in decision-making steps. A 10-point anchor scale from 0 (no effort was made) to 9 (every effort was made) with higher scores representing a greater perception of a shared decision-making effort.
HOBSCOTCH-CA fidelity as measured by CA participant's compliance with weekly homework assignments over the 8 weekly sessions. | At the beginning of HOBSCOTCH-CA (week 1) and at the end of the intervention (week 8).
  Homework assignments are given each week in which participants are asked to think about solutions using the Problem-Solving Therapy taught in the program. Compliance is measured by Yes (completed homework assignment) or No (did not complete homework assignment).
Changes in CA Participant Caregiver self-reported health status as measured by comparing scores on the Short-Form Health Survey 36 (SF-36) at baseline and 3 months-post intervention. | Baseline and 3 months post-intervention
  The Short Form Health Survey (SF-36) is a validated 36-item, patient- reported survey of patient health. It consists of 8 sub-scales, which are scored on a 3-point, 5-point or dichotomous (yes/no or true/false) scale. The scores are converted to a 1 - 100-point scale with a lower score indicating more disability, i.e. 0 = maximum disability and 100 = no disability.
Changes in CA Caregiver Participants' mood as measured by comparing scores on the Patient Health Questionnaire (PHQ-9) at baseline and at 3 months post- intervention. | Baseline and 3 months post-intervention
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria on a 4-point Likert scale as "0" (not at all) to "3" (nearly every day). Higher scores are consistent with greater symptoms of poor mood or depression.
Changes in CA Caregiver participants' anxiety as measured by comparing scores on the Generalized Anxiety Disorder-7 (GAD-7) at baseline and at 3-months post-intervention. | Baseline and 3 months post-intervention
  The Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring symptoms of generalized anxiety disorder (GAD). The seven items are scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Higher scores suggest greater symptoms of anxiety.
Changes in CA Participant Caregiver knowledge of relationship between their condition (brain cancer/tumor) and cognition and memory as measured by comparing scores on the HOBSCOTCH-CA Knowledge Questionnaire at baseline and at 6 months (end of study) | Baseline and at 6 months (end of study).
Feasibility of HOBSCOTCH-CA program for Caregivers as measured by study attrition and a Participant Satisfaction Survey. | At 6 months (end of study).
  The Participant Satisfaction Survey was developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It has been modified to address Caregiver's satisfaction as a result or participating in this study and contains 9 items scored on a 5- point Likert scale with a higher score indicating greater satisfaction with the program.
Sustainability of improvement on primary outcome measure of quality of life for Group 1 CA Participants by comparing scores on the Neuro-QOL at 3 months and 6 months post-intervention. | At 3 months and 6 months post-intervention
  The Neuro-QOL is a self-reported, validated assessment on health-related quality of life covering 17 domains in individuals with neurological disorders. Items are scored on a 5-point Likert scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. Depending on the domain, a higher or lower score can indicate better or poorer quality of life for that domain.
Sustainability of improvement on primary outcome measure of subjective cognition for Group 1 CA Participants by comparing scores on the Cognitive Function sub-scale of the Neuro-QOL at 3 months and 6 months post-intervention | At 3 months and 6 months post-intervention
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Sustainability of improvement on primary outcome measure of quality of life for Group 1 CA Participants by comparing scores on the FACT-Br at 3 months and 6 months post-intervention. | At 3 months and 6 months post-intervention
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is a validated instrument measuring general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 scales or domains. A 5-point Likert scale from 0 (not at all) to 4 (very much) is utilized with a higher score representing poorer or better QOL depending on the domain.
Sustainability of improvement on primary outcome measure for CA Participant Caregiver by comparing scores on the Zarit Caregiver Burden at 3 months and 6 months post-intervention. | At 3 months and 6 months post-intervention
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5 point Likert scale is used with a higher score indicating a greater level of perceived burden.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, MD, MPH, MSc, Principal Investigator — Dartmouth-Health/Dartmouth-Hitchcock, Dartmouth College
Locations (1):
- Dartmouth-Health Lebanon, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No